CLINICAL TRIAL: NCT03767790
Title: A Randomized Crossover Comparison of Model Predictive Control (MPC) Artificial Pancreas vs. Sensor Augmented Pump (SAP)/Predictive Low Glucose Suspend (PLGS) With Different Food Choices in the Outpatient Setting
Brief Title: Model Predictive Control (MPC) Artificial Pancreas vs. Sensor Augmented Pump (SAP)/Predictive Low Glucose Suspend (PLGS) With Different Food Choices in the Outpatient Setting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sansum Diabetes Research Institute (Other)
Collaborators: Harvard University (Other); Harvard School of Public Health (HSPH) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: G180011-S001
Record Dates: First submitted 2018-12-05; First posted 2018-12-07 (Actual); Last update posted 2019-08-08 (Actual); Status verified 2019-08

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: Artificial Pancreas; Hyperglycemia; Hypoglycemia; Nutrition
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Hyperglycemia; Hypoglycemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Automated Insulin Delivery (Experimental): Participants will use the Automated Insulin Delivery (AID) iAPS system for 2 weeks in the outpatient setting. During AID use, subjects will consume 6 study meals (3 meals of each meal type in assigned random order, 1-2 portions per meal,) at dinner time over the 2-week period in a pre-assigned random order, and document on the study meal forms when they consume each numbered meal.
  Interventions: Device: iAPS
- SAP/PLGS (No Intervention): Participants will use their home pump with a CGM sensor (sensor augmented pump) or in Predictive Low Glucose Suspend (PLGS) mode if their home pump supports this mode, for 2 weeks in the outpatient setting. During these 2 weeks, subjects will consume 6 study meals (3 meals of each meal type in assigned random order, 1-2 portions per meal,) at dinner time over the 2-week period in a pre-assigned random order, and document on the study meal forms when they consume each numbered meal.

INTERVENTIONS:
Device: iAPS — The AID system (iAPS) is comprised of an insulin pump, a Dexcom G6 continuous glucose monitoring sensor, and a smart phone that contains the algorithm and communicates with the other devices.
  Arms: Automated Insulin Delivery

SUMMARY:
The objective of this randomized crossover clinical trial is to 1) assess the efficacy and safety of an automated insulin delivery (AID) system using a Model Predictive Control (MPC) algorithm versus sensor augmented pump therapy (SAP)/Predictive Low Glucose Suspend (PLGS) in people with type 1 diabetes, and 2) assess the impact of different meal macronutrient content on glucose control when using AID and SAP.

DETAILED DESCRIPTION:
The goal of this study is to compare the efficacy and safety of an AID system using a MPC algorithm versus SAP/PLGS therapy with different food choices over a 4 week period.

The AID system (iAPS) is comprised of an insulin pump, a Dexcom G6 continuous glucose monitoring sensor, and a smart phone that contains the algorithm and communicates with the other devices.

In this study, during each two-week period, subjects will be given pre-weighed portions of different meals to eat (either regular semolina pasta or extra-long grain white rice) with detailed cooking instructions, and will eat these meals on 6 different occasions for dinner. They will bolus as they normally do for these meals. This will allow us to observe the postprandial meal response when using sensor-augmented pump (SAP) or iAPS, showing the importance of nutrition choices with modern technological treatments in T1D.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis, based on investigator assessment, of type 1 diabetes for at least one year and using insulin for at least 1 year.
* Using an insulin pump for at least 3 months at the time of screening. Insulin pump use includes use of automated features, to include predictive or threshold low-glucose suspend or hybrid closed-loop with without a Dexcom sensor.
* Familiarity and use of a carbohydrate ratio for meal boluses.
* Age ≥18.0 years old
* HbA1c < 10.5%, as performed by point of care or central laboratory testing. A1c will be assessed at the screening visit, or if already completed within 2 weeks of the screening visit, the prior lab value may be used in lieu of repeating this assessment.
* For females, not currently known to be pregnant. If female and sexually active, must agree to use a form of contraception to prevent pregnancy while a participant in the study. A negative serum or urine pregnancy test will be required for all females of child-bearing potential. Participants who become pregnant will be discontinued from the study. Also, participants who during the study develop and express the intention to become pregnant within the timespan of the study will be discontinued.
* Willingness to switch home pump to PLGS or full manual mode if using hybrid closed-loop with an FDA approved system.
* Have an emergency contact living at home with the subject who will be available to be contacted by the study staff overnight in the event of an emergency.
* Investigator has confidence that the participant can successfully operate all study devices and is capable of adhering to the protocol, to include having basic cooking equipment at home to prepare the study meals.
* Willingness to switch to lispro (Humalog) or aspart (Novolog) if not using already, and to use no other insulin besides lispro (Humalog) or aspart (Novolog) during the study.
* Willingness not to start any new non-insulin glucose-lowering agent during the course of the trial.

Exclusion Criteria:

* Use of an unapproved closed-loop insulin delivery system within 2 weeks before screening or during the study is not allowed.
* Gastrointestinal disease such as celiac disease or multiple food allergies.
* Any form of gluten sensitivity or wheat allergy.
* Allergies to any form of nuts or ingredients present in the study meals (tomatoes etc).
* History of difficulty digesting food.
* Concurrent use of Afrezza or any non-insulin glucose-lowering agent other than metformin (including GLP-1 agonists, Symlin, DPP-4 inhibitors, SGLT-2 inhibitors, sulfonylureas).
* Hemophilia or any other bleeding disorder
* One or more episodes of hypoglycemia requiring an emergency room visit or hospitalization in the past 6 months.
* One or more episodes of hyperglycemia requiring an emergency room visit or hospitalization in the past 6 months.
* Self-reported or clinically documented hypoglycemia unawareness.
* A condition, which in the opinion of the investigator or designee, would put the participant or study at risk
* Participation in another pharmaceutical or device trial at the time of enrollment or during the study
* Having a direct supervisor at place of employment who is also directly involved in conducting the clinical trial (as a study investigator, coordinator, etc.); or having a first-degree relative who is directly involved in conducting the clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-01-03 (Actual); Primary Completion 2019-06-27 (Actual); Study Completion 2019-06-27 (Actual)

PRIMARY OUTCOMES:
Time in target glucose range | 4 weeks
  Time in target glucose range 70-180 mg/dL measured by CGM to determine safety and efficacy of the integrated system

SECONDARY OUTCOMES:
Postprandial glucose peak | 4 weeks
  Postprandial glucose peak rise (highest measurement in mg/dL) from baseline glucose (mg/dl) for the 5-hour period after the study meals, during both use of SAP/PLGS and when using the iAPS
Time to postprandial glucose peak | 4 weeks
  Time (minutes) to postprandial glucose (highest measurement in mg/dL) rise from baseline glucose (mg/dl) during the 5-hour period after the study meals, during both use of SAP/PLGS and when using the iAPS
Postprandial Area Under the Curve | 4 weeks
  Area Under the Curve Glucose (mg/dl x min) for the 5-hour period after the study meals, during both use of SAP/PLGS and when using the iAPS
Postprandial time for glucose to return to baseline | 4 weeks
  Time (minutes) for CGM glucose to return to baseline (starting value) after the study meals, during both use of SAP/PLGS and when using the iAPS
Glucose < 70 mg/dL | 4 weeks
  Percent time GGM glucose < 70 mg/dL
Glucose < 54 mg/dL | 4 weeks
  Percent time GGM glucose < 54 mg/dL
Glucose > 180 mg/dL | 4 weeks
  Percent time GGM glucose > 180 mg/dL
Glucose > 250 mg/dL | 4 weeks
  Percent time GGM glucose > 250 mg/dL
Serious adverse events (SAE) | 4 weeks
  The total number of serious adverse events during the clinical trial
Serious adverse device events (SADE) | 4 weeks
  The total number of serious adverse events related to the study device use during the clinical trial
Adverse device effects (ADE) | 4 weeks
  The total number of adverse device effects (ADE) during the clinical trial
Unanticipated adverse device effects (UADE) | 4 weeks
  The total number of unanticipated adverse device effects (UADE) during the clinical trial

OTHER OUTCOMES:
Total daily insulin use | 4 weeks
  Total daily insulin use (units/day) during both use of SAP/PLGS and when using the iAPS
Total basal insulin use | 4 weeks
  Total daily basal insulin use (units/day) during both use of SAP/PLGS and when using the iAPS
Total bolus insulin use | 4 weeks
  Total daily bolus insulin use (units/day) during both use of SAP/PLGS and when using the iAPS
Sensor Use Time | 4 weeks
  Total hours of CGM sensor use time during both use of SAP/PLGS and when using the iAPS
Closed-Loop Active Time | 2 weeks
  Percent time (hours/day) of closed-loop use during the two weeks of iAPS use
Device Issues | 4 weeks
  Total number of devices issues during the clinical trial

CONTACTS AND LOCATIONS:
Overall Officials: Eyal Dassau, PhD, Principal Investigator — John A. Paulson School of Engineering and Applied Sciences; David Eisenberg, MD, Principal Investigator — Harvard School of Public Health (HSPH); Jordan E Pinsker, MD, Principal Investigator — Sansum Diabetes Research Institute
Locations (1):
- Sansum Diabetes Research Institute, Santa Barbara, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Deshpande S, Pinsker JE, Church MM, Piper M, Andre C, Massa J, Doyle Iii FJ, Eisenberg DM, Dassau E. Randomized Crossover Comparison of Automated Insulin Delivery Versus Conventional Therapy Using an Unlocked Smartphone with Scheduled Pasta and Rice Meal Challenges in the Outpatient Setting. Diabetes Technol Ther. 2020 Dec;22(12):865-874. doi: 10.1089/dia.2020.0022. Epub 2020 Oct 13. PMID 32319791